CLINICAL TRIAL: NCT02969928
Title: Full-mouth Periodontal Debridement Associated With Two Different Antibiotic Agents to Treat Generalized Aggressive Periodontitis: Randomized Controlled Clinical Trial
Brief Title: Two Different Antibiotic Agents to Treat Generalized Aggressive Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AmxMetClmCFA
Record Dates: First submitted 2016-11-07; First posted 2016-11-21 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Aggressive Periodontitis
Keywords: Full-mouth ultrasonic debridement; Clarithromycin; Amoxicillin; Metronidazole
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Periodontal Debridement; Clarithromycin; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin and Metronidazole (Active Comparator): In this group (n = 23), patients will take Amoxicillin 500 mg tid for 7 days and Metronidazole 400 mg tid for 7 days and full-mouth ultrasonic debridement will be performed to treat diseased sites.
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Amoxicillin; Drug: Metronidazole
- Clarithromycin (Experimental): In this group (n = 23), patients will take Clarithromycin 500 mg bid for 7 days and full-mouth ultrasonic debridement will be performed to treat diseased sites.
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Clarithromycin

INTERVENTIONS:
Procedure: Full-mouth ultrasonic debridement — Full-mouth ultrasonic debridement will be performed in order to treat diseased sites
  Other Names: Periodontal debridement
Drug: Clarithromycin — Administration of Clarithromycin 500mg bid for 7 days
  Other Names: Biaxin
  Arms: Clarithromycin
Drug: Amoxicillin — Administration of Amoxicillin 500mg tid for 7 days.
  Other Names: Amoxil
  Arms: Amoxicillin and Metronidazole
Drug: Metronidazole — Administration of Metronidazole 400mg tid for 7 days.
  Other Names: Flagyl
  Arms: Amoxicillin and Metronidazole

SUMMARY:
The aim of this study is to assess the clinical outcomes of full-mouth ultrasonic debridement combined with clarithromycin or amoxicillin + metronidazole association for the treatment of generalized aggressive periodontitis (GAgP).

DETAILED DESCRIPTION:
The study methodology is according to CONSORT-STATEMENT 2010 for randomized controlled clinical trials.

Study Design

The study is designed as a prospective, interventional, parallel, triple blind, randomized, controlled clinical trial aimed to assess the clinical outcomes of full-mouth ultrasonic debridement combined with clarithromycin or amoxicillin + metronidazole association for the treatment of generalized aggressive periodontitis (GAgP). The study was approved by Institute of Science and Technology's (ICT - State University of São Paulo) Ethics Committee (protocol 1.079.307).

Source of data

The population of this study will be recruited among patients referred to the Science and Technology Institute - ICT- São José dos Campos, College of Dentistry. Patients will fill a healthy history questionnaire to ensure that they are medically qualified for participate in this study. Based on the power calculation for this study, 44 subjects divided into two groups will be needed to achieve 80% power to detect a 0.8 mm difference in the clinical attachment level (CAL) of patients.

Clinical Parameters

All clinical parameters will be assessed by a single blinded, trained and calibrated examiner (CFA) before periodontal therapy (baseline) and at 3 and 6 months after using a manual probe. Measurements will be done at six sites per tooth (mesiobuccal, buccal, disto-buccal, distolingual, lingual, and mesiolingual) in all teeth, except third molars.

The following clinical parameters will be evaluated: 1) Full-mouth plaque index (FMPI); 2) Bleeding on probing (BoP); 3) Probing depth (PD): distance from the bottom of sulcus/pocket to gingival margin; 4) Gingival recession (GM): distance from the free gingival margin to cement-enamel junction (CEJ); 5) Clinical attachment level (CAL): distance from bottom of sulcus/pocket to the CEJ. The CEJ will be identified by careful probe on cervical area.

Calibration and Randomization

Initially, a total of ten patients presenting with GAgP will be selected. The designated examiner (CFA) will measure CAL and PD in all patients twice within 24 hours, with an interval of ≥ 1 hour between examinations. Then, the measures will be submitted to intraclass correlation test and the examiner will be judged calibrated if reaches 90% agreement.

Patients will be allocated into two groups according to a computer-generated list. The allocation will be implemented by an investigator (NCCS) who was not directly involved in the examination or treatment procedures. All medication will be prepared and encased in identical opaque coded bottles by a manipulation pharmacy on São José dos Campos/São Paulo.

Treatment Protocols

All patients will be treated with periodontal therapy through of the one-stage, full mouth, ultrasonic debridement (FMUD). In a single session, patients will receive local anesthesia and periodontal debridement with ultrasound equipment (Cavitron - Dentsply EUA) and subgingival tips (UI25KSF10S, Hu-Friedy). All diseased sites will be instrumented in this one session. The debridement session will be performed by a single experienced and trained periodontist (MPS), different from the examiner. Immediately before the mechanical therapy, patients will be allocated in one of the two treatment protocols:

1. Clarithromycin (CLM) group (n = 22): FMUD + CLM 500 mg bid, for 7 days and
2. Amoxicillin (AMX) + metronidazole (MET) group (n = 22): FMUD + (AMX 500 mg tid + MET 400 mg tid, both for 7 days.

All patients will start taking the pills immediately before of the FMUD session.

Compliance and Adverse Effects

After 7 days of periodontal treatment, patients will be asked to return any medication not taken and/or the empty bottles. The number of pills not taken by the subject will be documented. Moreover, patients will be instructed to return a self-report form filled about any possible adverse effects in order to help evaluate their adherence to the systemic antimicrobial regimen.

Statistical analysis

Mean and standard deviation will be calculated for each parameter. The normal distribution of the data will be analyzed by Shapiro-Wilk test. Data from clinical measurements will be subjected to analysis of variance (repeated measures) for inter and intra-group comparison.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of GAgP (AAP, 1999);
2. presence of ≥20 teeth;
3. presence of ≥ 6 sites presenting PD ≥ 5mm with bleeding on probing (BOP) and ≥2 sites with PD ≥7mm (including incisors and first molars, in addition to other two non-contiguous teeth);
4. good general health;
5. ≤ 35 years old; and
6. agree to participate in the study and sign a written informed consent. All subjects will be individually informed about the objectives, probable risks and benefits of the protocol treatment (according to Resolution nº196 of October 1996 and to the Professional Code of Dental Ethics - 179/93).

Exclusion Criteria:

1. pregnancy or lactating;
2. suffer from any systemic disease (e.g. cardiovascular disorders, diabetes, blood dyscrasias, immunodeficiency, etc) which could alter the course of periodontal disease;
3. took antimicrobials in the previous 6 months;
4. taking long-term anti-inflammatory drugs;
5. previous periodontal treatment within the last 12 months;
6. smokers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- College of Dentistry - São José dos Campos, Sao Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradeep AR, Kathariya R. Clarithromycin, as an adjunct to non surgical periodontal therapy for chronic periodontitis: a double blinded, placebo controlled, randomized clinical trial. Arch Oral Biol. 2011 Oct;56(10):1112-9. doi: 10.1016/j.archoralbio.2011.03.021. Epub 2011 May 6. PMID 21529775
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Duarte PM, Lira EA, Faveri M. Short-term benefits of the adjunctive use of metronidazole plus amoxicillin in the microbial profile and in the clinical parameters of subjects with generalized aggressive periodontitis. J Clin Periodontol. 2010 Apr;37(4):353-65. doi: 10.1111/j.1600-051X.2010.01538.x. PMID 20447259
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Derived] Araujo CF, Andere NMRB, Castro Dos Santos NC, Mathias-Santamaria IF, Reis AA, de Oliveira LD, Jardini MAN, Casarin RCV, Santamaria MP. Two different antibiotic protocols as adjuncts to one-stage full-mouth ultrasonic debridement to treat generalized aggressive periodontitis: A pilot randomized controlled clinical trial. J Periodontol. 2019 Dec;90(12):1431-1440. doi: 10.1002/JPER.18-0399. Epub 2019 Jul 16. PMID 31257591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: Evaluate the difference between baseline and 6 months CAL measures.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Number analyzed (Participants) | 23 | 23
mm
  Baseline | 3.69 (0.7) | 3.62 (0.4)
  3 months | 2.4 (0.5) | 3 (0.4)
  6 months | 3 (0.5) | 3 (0.4)

2. Secondary Outcome: Change in Probing Depth (PB)
Description: Evaluate the difference between baseline and 6 months PB measures.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Number analyzed (Participants) | 23 | 23
mm
  Baseline | 3.44 (0.6) | 3.41 (0.4)
  3 months | 2.5 (0.3) | 2.7 (0.2)
  6 months | 2.6 (0.3) | 2.7 (0.25)

3. Secondary Outcome: Change in Bleeding on Probe (BoP)
Description: Evaluate the difference between baseline and 6 months BoP measures.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: % of sites with bleeding on probe
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Number analyzed (Participants) | 23 | 23
% of sites with bleeding on probe
  Baseline | 53.4 (17.4) | 43.7 (8.3)
  3 months | 30.2 (9.3) | 24.8 (9.8)
  6 months | 27.3 (8.3) | 23.3 (9.3)

4. Other Pre Specified Outcome: Compliance
Description: After 7 days of periodontal treatment, patients will be asked to return any medication not taken and/or the empty bottles. The number of pills not taken by the subject will be documented in order to evaluate compliance.
Time Frame: One week post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Number analyzed (Participants) | 23 | 23
Participants
  # of patients that did not take ≥1 pills | 3 | 4
  # of patients that interrupted the drug intake | 2 | 0

5. Other Pre Specified Outcome: Adverse Effects That May be Related to Antibiotic Treatment
Description: Patients will be instructed to fill a self-report form about any possible adverse effects in order to help evaluate their adherence to the systemic antimicrobial regimen.
Time Frame: One week post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
Number analyzed (Participants) | 23 | 23
Participants
  Headache | 1 | 2
  Stomach pain | 4 | 3
  Nausea/vomiting | 3 | 6
  Metallic taste | 7 | 13
  Diarrhea/abdominal pain | 3 | 3
  Drowsiness | 2 | 3
  Itching | 1 | 0
  Skin wounds | 0 | 0
  None | 5 | 5

ADVERSE EVENTS:
Time Frame: during 7 days post-treatment
Description: 7 days after the therapy patients returned to fill out a self-report form about 8 possible adverse effects resulting from the antibiotic intake, based on Martys: Headache, Stomach pain, Nausea/vomiting, Metallic taste, Diarrhea/ abdominal pain, Drowsiness, Itching and Skin wounds.
Arm/Group | Amoxicillin and Metronidazole | Clarithromycin
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 18/23 | 18/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amoxicillin and Metronidazole (N=23) | Clarithromycin (N=23)
Headache (General disorders) | 1 | 2
Stomach pain (Gastrointestinal disorders) | 4 | 3
Nausea/vomiting (General disorders) | 3 | 6
Metallic taste (General disorders) | 7 | 13
Diarrhea/ abdominal pain (Gastrointestinal disorders) | 3 | 3
Drowsiness (General disorders) | 2 | 3
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Skin wounds (Skin and subcutaneous tissue disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No